CLINICAL TRIAL: NCT03810924
Title: Stress-related Predictor Profiles for Craving and Relapse in Human Addiction
Brief Title: Stress-related Predictor Profiles in Human Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Project Group for Automation in Medicine and Biotechnology PAMB, Mannheim (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRR265 A03
Record Dates: First submitted 2018-11-26; First posted 2019-01-22 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Alcohol Use Disorder; Stress Reaction; Social Stress; Craving; Relapse; Addiction; Risk Behavior
MeSH Terms: conditions — Alcoholism; Fractures, Stress; Recurrence; Behavior, Addictive; Risk-Taking | interventions — Psychological Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Participants reads newspaper before Barlab-Exposure
  Interventions: Behavioral: Barlab-Exposure; Behavioral: Reading Newspaper
- Experimental 1 (Distress) (Experimental): Participants undergo the Trier Social Stress Test before Barlab-Exposure
  Interventions: Behavioral: Trier Social Stress Test; Behavioral: Barlab-Exposure
- Experimental 2 (Eustress) (Experimental): Participants ride an ergometer before Barlab-Exposure
  Interventions: Behavioral: Ergometer; Behavioral: Barlab-Exposure

INTERVENTIONS:
Behavioral: Trier Social Stress Test — Test to induce high levels of acute social stress, including actors and a faked exam situation
  Arms: Experimental 1 (Distress)
Behavioral: Ergometer — Riding ergometer
  Arms: Experimental 2 (Eustress)
Behavioral: Barlab-Exposure — Participants are exposed to a bar situation with different sorts of alcohol available. They sniff at water and at one alcoholic drink.
Behavioral: Reading Newspaper — Participants read newspaper
  Arms: Control

SUMMARY:
Long-term aim is the definition of a setup of mobile sensors and their integration in a mobile infrastructure that allows the prediction of stress related alcohol intake in an ambulatory setting. Here, we aim to identify stress- and alcohol cue-related physiological markers in a lab experiment to assess interactions between acute psychological vs. physical stress exposure and alcohol cue-exposure regarding their effects on measures relevant for the development and maintenance of Alcohol Use Disorder (AUD). Further, we aim to identify neural correlates in brain circuits of motivational, cognitive, and affective processing. In addition to applying established stress-related markers, we will integrate innovative sensor-based measures.

DETAILED DESCRIPTION:
In patients with Alcohol Use Disorder (AUD) stress exposure is known to affect craving, cue-reactivity and relapse risk. Here, we aim to identify stress- and alcohol cue-related physiological markers in a lab experiment to assess interactions between acute psychological vs. physical stress exposure and alcohol cue-exposure regarding their effects on (1) alcohol craving and related markers (attentional bias to alcohol-cues, implicit association task, neural cue-reactivity), (2) their predictive capacity for future alcohol intake, (3) the identification their neural correlates in brain circuits of motivational, cognitive, and affective processing. In addition to applying established stress-related markers (cortisol in saliva, heart-rate variability, systolic blood pressure and electrodermal activity), (4) we will integrate portable sensors (wearables) to allow a future integration in ambulatory assessments and to test innovative measures currently under investigation (e.g. voice stress analysis) to identify whether these additional parameters increase the predictive significance. Our long-term aim is the definition of a setup of mobile sensors and their integration in a mobile infrastructure that allows the prediction of stress related alcohol intake in an ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol-use disorder according to 2 DSM-V criteria not requiring detoxification: AUD subjects with mild AUD will fulfill at least 2 and not more than 5 diagnostic criteria; a second group of AUD subjects will fulfill 4-5 criteria for moderate AUD
* sufficient ability to communicate with the investigators, to answer questions in oral and written form
* fully informed consent
* written informed consent

Exclusion Criteria:

* withdrawal of the declaration of consent
* Pregnancy
* Using hormonal contraceptives
* Perimenopausal/ postmenopausal
* positive urin drug screening (cannabis, amphetamine, opiates, benzodiazepines, cocaine)
* Lifetime history of DSM-5 bipolar disorder, schizophrenia or schizophrenia spectrum disorder, or substance dependence other than alcohol or nicotine or cannabis dependence.
* Current threshold DSM-5 diagnosis of major depressive disorder, or presence of suicidal intention
* History of severe head trauma or other severe central nervous system disorder (e.g., dementia, Parkinson's disease, multiple sclerosis)
* Current use of medications or drugs known to interact with the CNS within at least four half-lives post last intake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
change in heart rate | at examination day: continuous measurement throughout the whole experiment (except during MRI scanning); duration around 2 hours; starting 1 hour 50 minutes after arrival of the proband
  heart rate acquired with ear clip (continuous time series)
change in heart rate variability | at examination day: continuous measurement throughout the whole experiment (except during MRI scanning); duration around 2 hour; starting 1 hour 50 minutes after arrival of the proband
  heart rate variability acquired with ear clip (continuous time series)
change in blood pressure (systolic and diastolic) | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at hours:minutes 2:20, 2:50, 3:20, 3:50, 4:50, 5:05 after arrival of the proband
  acquired with pressure sleeve
change in electrodermal activity | at examination day: continuous measurement throughout the whole experiment (except during MRI scanning); duration around 2 hour; starting 1h 50min after arrival of the proband
  time series acquired with body sensor
neural alcohol-related cue-reactivity | at examination day: measured directly after the behavioral tasks at the end of the lab experiment
  % signal change, measured with fMRI; paradigm Vollstädt-Klein et al. 2010; [% signal change is not a change over time; it is measured during one experimental session]
neural inhibition processing | at examination day: measured directly after the behavioral tasks at the end of the lab experiment
  % signal change, measured with fMRI; stop-signal reaction time task (Fauth-Buhler et al. 2012) [% signal change is not a change over time; it is measured during one experimental session]
neural emotion processing | at examination day: measured directly after the behavioral tasks at the end of the lab experiment
  % signal change, measured with fMRI; faces task (Hariri et al. 2002) [% signal change is not a change over time; it is measured during one experimental session]
resting state activity | at examination day: measured directly after the behavioral tasks at the end of the lab experiment
  resting state connectivity measured with fMRI
fMRI | at examination day: measured directly after the behavioral tasks at the end of the lab experiment
  neural alcohol-related cue-reactivity, stop-signal reaction time task, emotion processing and resting state fMRI
attentional bias to alcohol cues | at examination day: measured directly after the stress task / newspaper reading; before "implicit alcohol association" and MRI session
  measured with reaction time differences (in milliseconds) using the dotprobe-task (Vollstädt-Klein et al. 2009) [reaction time differences is not a change over time; it is measured during one experimental session]
implicit alcohol association | at examination day: measured after the stress task / newspaper reading, directly after the "attentional bias to alcohol cues" ; before MRI session
  measured with reaction time differences (in milliseconds) using the implicit association task (Wiers et al. 2016) [reaction time differences is not a change over time; it is measured during one experimental session]
change in level of cortisol | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at hours:minutes 2:20, 2:50, 3:20, 3:50, 4:50, 5:05 after arrival of the proband
  cortisol measured in saliva as a stress marker
change in voice stress pattern | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at hours:minutes 2:20, 2:50, 3:20, 3:50, 4:50, 5:05 after arrival of the proband
  audio file of participants' voice for voice stress pattern analysis will be recorded. From this a multivariate measure (i.e. multivariate vector) will be acquired (including frequency, loudness etc.)
change in alcohol urges | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at hours:minutes 2:20, 2:50, 3:20, 3:50, 4:50, 5:05 after arrival of the proband
  self-report questionnaire: "Alcohol Urge Questionnaire (AUQ)"; Bohn et al. 1995
change in alcohol craving | at examination day: 6 time points measured throughout the whole experiment (except during MRI scanning); at hours:minutes 2:20, 2:50, 3:20, 3:50, 4:50, 5:05 after arrival of the proband
  self-report "How strong is your craving for alcohol?": reported on a visual analogue scale ranging from 0 to 100

SECONDARY OUTCOMES:
alcohol consumption | 12 months follow-up
  self-report using the instrument Form90 (Scheurich et al. 2005)

CONTACTS AND LOCATIONS:
Overall Officials: Falk Kiefer, Prof., Principal Investigator — Central Institute of Mental Health, Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No